CLINICAL TRIAL: NCT06043167
Title: Clinimetric Application of FOUR Scale as in Treatment and Rehabilitation of Patients With Acute Cerebral Injury. - a Prospective Observational Mono-center Cohort Study
Brief Title: Clinimetric Application of FOUR Scale as in Treatment and Rehabilitation of Patients With Acute Cerebral Injury
Acronym: FOURACI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Surgut Clinical Trauma Hospital (Other)
Collaborators: Ural State Medical University (Other)
Responsible Party: Principal Investigator, Andrey Belkin, MDRussian Federation of Anesthesiologists and Reanimatologists, Ural State Medical University
Other Study IDs: 523721
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Acute Traumatic Brain Injury; Subarachnoid Hemorrhage
MeSH Terms: conditions — Stroke; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The predictive value russian rendition the FOUR score. — It is planned to include at least 200 adult OAR patients and all those transferred to the rehabilitation department for evaluation.
  To maintain accounting documentation, an individual registration card is offered for registration. The paper version of the IRC records the age of the patient, the diagnosis according to the International Classification of diseases of the tenth revision (ICD-10), the day of hospital stay and ICU. The level of consciousness is assessed according to the unified interdisciplinary scale of disorders of consciousness, Glasgow Coma Scale (GCS), Full Outline of Unresponsiveness (FOUR) and Richmond Agitation-Sedation Scale (RASS). After each inspection, the data is entered into the electronic version of the IRC.

SUMMARY:
The aim of this study is to increase the effectiveness of clinical monitoring of patients with acute cerebral insufficiency by improving the discriminative ability of the FOUR scale. To study the sensitivity and specificity of the FOUR scale as a clinimetric of chronic disorders of consciousness.

DETAILED DESCRIPTION:
The key step in choosing a strategy for treating acute cerebral insufficiency is the assessment of the severity of cerebral damage and prognosis. The importance of correcting the severity of damage and prognosis for the choice of treatment strategy is beyond doubt.

At the same time, the complexity of objective evaluation is preserved throughout the world, after more than 40 years, has become an integral part of clinical practice worldwide. The findings obtained using GCS showed a strong relationship with those obtained using other indicators of severity and outcome. Although the scale of Glasgow coma is considered routine method, it has a number of significant drawbacks.

First, the verbal response of GCS tests often becomes inadequate in psychomotor-excited patients. On the contrary, in many patients with depressed consciousness, the verbal response is insufficient. Moreover, the GSC verbal response assessment cannot be applied to critical patients or those who have undergone intubation.

Secondly, and most importantly, GSC does not assess brain stem reflexes, eye movements, or complex motor responses in patients with altered consciousness. In addition, the GCS score is numerically skewed toward the motor response (the maximum number of points given for the motor response). These deficiencies previously caused repeated attempts to improve GCS: reaction level scale (RLS85), comprehensive consciousness level Scale (CLOCS), clinical neurological assessment (CNA) , Coma Recovery Scale (CRS), Glasgow-Liege Scale (GLS), Innsbruck Coma Scale (ICS), 15 and 60-second test (SST). Similar scans, tests are very long and laborious. None of these subsequently gained enough weight to replace GCS.

Third, despite the fact that GSC is regularly used in therapeutic and surgical intensive care units and resuscitation units, as well as the fact that it is usually used in conjunction with the APACHE system assessment, reliability in predicting outcomes in patients is unsatisfactory. Fourthly, Rowley and Fielding found that the reliability of the GCS score increases with the experience of its users and that user inexperience is associated with a high error rate.

The new coma scale, Full Outline of UnResponsiveness (FOUR), is based on the minimum number of tests needed to analyze the severity of cerebral damage and prognosis. Universal and suitable, including for patients with altered consciousness. The FOUR scale has four categories studied. In contrast to GCS, the number of components and the maximum rating in each category are four (E4, M4, B4, R4). This is significantly easier than in GCS with different points for each category. The FOUR scale is suitable for assessing a patient with a locked person syndrome, as well as in the presence of a vegetative state. Conditions when the eyes can open spontaneously, but cannot follow the pointer. The motor or motor component is recorded primarily on the limb. Response options include the presence of status epilepticus, myoclonus. Also, the motor response combines decorticative regimen and generalized myoclinic status. Hand position tests (thumb up, fist, and peace sign) are reliable for assessing wakefulness. Three reflexes assessing brain stem depression, testing the functions of the midbrain, pons and medulla oblongata, are used in various combinations. The clinical sign of acute dysfunction of the third pair of FMN (unilateral pupil dilation), pupillary and oculomotor reactions is assessed. Separately, the functioning of the respiratory center, as the lower part of the brain stem, is considered. In intubated patients, the presence of independent attempts between cycles of mechanical ventilation is assessed. The value of 0 in all responses is the basis for considering the diagnosis of brain death. The FOUR evaluation of the lung is reproducible and takes several minutes.

In order to increase the effectiveness of clinical monitoring of patients with acute cerebral insufficiency by improving the discriminatory ability of the FOUR scale, and to study the sensitivity and specificity of the scale as clinimetrics of chronic disorders of consciousness, a study was initiated: Clinimetric application of FOUR scale as in treatment and rehabilitation of patients with Acute Cerebral Injury - FOURACI.

The aim of this study is to increase the effectiveness of clinical monitoring of patients with acute cerebral insufficiency by improving the discriminative ability of the FOUR scale. To study the sensitivity and specificity of the FOUR scale as a clinimetric of chronic disorders of consciousness.

A monocenter prospective non-randomized cohort study is planned using a continuous sampling method on the basis of the Surgut Clinical Trauma Hospital of the Khanty-Mansiysk Autonomous Okrug - Yugra in the department of anesthesiology - intensive care, ICU for patients with chronic impaired consciousness and the department of medical rehabilitation of patients with CNS disorders.

The objectives of the study are:

1. To investigate the sensitivity of FOUR in the range of values <8 to the dynamics of the state in comparison with the GCS scale and the unified interdisciplinary scale of disorders of consciousness (A.N.Konovalova).
2. Stratify the ranges of values of the FOUR scale from the position of outcomes according to GOS and PITC in ICU patients with different resuscitation syndromes.
3. Calibrate the FOUR scale to assess the prognosis of the outcome of the course of the OCN in the acute (in ICU patients) and subacute (rehabilitation department) period.

It is planned to include at least 200 adult OAR patients and all those transferred to the rehabilitation department for evaluation.

To maintain accounting documentation, an individual registration card is offered for registration. The paper version of the IRC records the age of the patient, the diagnosis according to the International Classification of diseases of the tenth revision (ICD-10), the day of hospital stay and ICU. The level of consciousness is assessed according to the unified interdisciplinary scale of disorders of consciousness, Glasgow Coma Scale (GCS), Full Outline of Unresponsiveness (FOUR) and Richmond Agitation-Sedation Scale (RASS). The severity of the patient's condition is assessed according to the scales: comorbidity Index, Behavior Pain Assessment (BPS), Acute Physiology and Chronic Health Evaluation II (APACHE II), Sepsis-related Organ Failure Assessment (SOFA), Glasgow Outcome Scale (GOS). After each inspection, the data is entered into the electronic version of the IRC.

ELIGIBILITY:
Inclusion Criteria:

* acute brain failure after stroke or acute brain trauma

Exclusion Criteria:

* the inability to assess the factors included in the study.
* cardiopulmonaryresuscitation
* arterial hypotension
* hypoxemia
* malignant hyperthermia or hypothermia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult atients with syndrome of acute cerebral insufficiency
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
The interrater reliability of russian rendition the FOUR score | 2023 - 2024

OTHER OUTCOMES:
The predictive value russian rendition the FOUR score. | 2023 - 2024

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Belkin, Principal Investigator — Russian Federation of Anesthesiologists and Reanimatologists
Locations (1):
- Surgut Clinical Trauma Hospital, Surgut, Khanty-Mansi Autonomous Okrug - Yugra, Russia

IPD SHARING:
Plan to Share IPD: No